CLINICAL TRIAL: NCT02771873
Title: A Family Based Randomized Controlled Trial of Cardiovascular Risk Reduction in Individuals With Family History of Premature Coronary Heart Disease in India
Brief Title: Programme of Lifestyle Intervention in Families for Cardiovascular Risk Reduction
Acronym: PROLIFIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health Foundation of India (Other)
Collaborators: Sree Chitra Tirunal Institute for Medical Sciences & Technology (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LN0181
Record Dates: First submitted 2016-05-05; First posted 2016-05-13 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual care (No Intervention): Screening for CVD risk factors plus one time education regarding management of risk factors will be provided to all family members.
- Life style Intervention and care coordination (Experimental): Integrated cardiovascular disease risk management.
  Interventions: Behavioral: Integrated cardiovascular disease risk management.

INTERVENTIONS:
Behavioral: Integrated cardiovascular disease risk management. — Health promotion intervention
  Arms: Life style Intervention and care coordination

SUMMARY:
The overall goal of the study is to test the effectiveness and sustainability of an integrated care model for managing cardiovascular risk in individuals with family history of premature coronary heart disease (CHD).

This care model involves:

1. screening for cardiovascular risk factors,
2. providing lifestyle interventions for prevention and management of cardiovascular risk factors,
3. providing a framework for linkage to appropriate primary health care facility and
4. active follow-up of intervention adherence.

Initially, a formative qualitative research component will gather information on understanding of diseases, barriers to care, specific components of the intervention package (for example, context specific ways to enhance physical activity and to reduce prolonged sitting time, ways to improve diet etc.) and feedback on the intervention strategies (lifestyle education, care and linkage coordination). Then a randomized controlled trial involving ~700 families and 1400 participants will be used to determine whether an integrated care model is effective in reducing or halting the progression of CHD risk factors and risk factor clustering in families. The sustainability and scalability of this intervention will be assessed through economic and qualitative lenses to estimate value and acceptability. Scalability will be informed by cost-effectiveness and acceptability of the integrated cardiovascular risk reduction approach.

DETAILED DESCRIPTION:
STUDY AIMS:

AIM 1. To identify barriers to implementing an integrated cardiovascular risk management program in families of individuals with a positive history CHD.

AIM 2. To assess the effectiveness of an integrated cardiovascular risk management strategy (consisting of screening for risk factors, lifestyle education and linkage to primary care for cardiovascular risk factor management) on risk factor clustering in families, and changes in blood pressure (BP), lipids, glucose, smoking and physical activity.

AIM 3. To estimate the scalability of the integrated cardiovascular risk reduction strategy in families of individuals with a positive history CHD for state- or nation-wide implementation. Scalability will be informed by cost-effectiveness and acceptability of the integrated cardiovascular risk reduction approach.

STUDY DESIGN:

The proposed project uses mixed methods to achieve the study aims, the three design approaches include:

Aim 1, formative qualitative research; Aim 2, a randomized controlled trial; and Aim 3, cost effectiveness and evaluative qualitative research.

Additionally a pilot study will be conducted with the aim to understand the practical feasibility of the study, acceptability among participants, appropriateness of the study tools and finally to explore the interests of other stakeholders (community health workers and department of health service, Government of Kerala). The pilot study will include only 30 participants. It is essentially to check the validity of the responses elicited from the tools. We also plan to conduct two focus group discussions with the potential participants (individuals with family history of CHD). Additionally, 6 in-depth interviews will be conducted with community health workers (convenient sampling) to assess their opinion about the intervention programme.

Formative qualitative research (Aim 1):

Semi-structured focus group discussions (FGDs) of 6-12 adults with family history of CHD will gather information on understanding of diseases, barriers to care, and feedback on the intervention (lifestyle education, care and linkage coordination). In-depth interviews with stake-holders (frontline community health care workers (FCHW), primary care physicians, and general practitioners) will be face-to-face and semi-structured and will include questions regarding integration of cardiovascular risk management at the family level. The intervention and trial protocols will be modified to incorporate key findings collected from FGDs and interviews to make the intervention more contextually-relevant.

Integrated cardiovascular risk reduction intervention (Aim 2):

A randomized controlled trial of families of individuals with a positive history CHD will be used to address Aim 2. Eligibility criteria: Eligible families include those with at least one family member with physician confirmed CHD diagnosed before the age of 55 years. If there are family members who have died from CHD (physician confirmed deaths) before the age of 55 years, such families will be also eligible to participate in the study. The medical records of CHD patients will be used to confirm the diagnosis and the age of the index case. A written informed consent to the study randomization plan from the head of the family is a mandatory eligibility criteria. All participating family members will also be required to provide individual consent to participate. Family randomization: Each family will randomly be assigned to participate in either the treatment intervention arm (integrated CVD risk management) or usual care arm (no interventions other than initial screening). Participants eligibility criteria: Minimum of two members from each family will be included even if they reside in separate houses. Potential participants must be either parents, children or brothers and sisters of the affected person (individual with history of CHD) in order to enter the study and more than 18 years of age.

Bedridden and terminally ill patients will be excluded from the study.

To address Aim 2, several clinical outcomes will be assessed. Primary outcome: proportions in each group achieving or improving risk factor control status (blood pressure<140/90 mmHg, fasting blood glucose (FPG)<110 mg/dl, low-density lipoprotein (LDL)<100 mg/dl, abstinence from smoking/tobacco use: at least 3 out of 4 risk factors).

Secondary outcomes:

1. between group difference in number of optimal CV health indicators (BP<120/80 mmHg, TC<200 mg/dl, FPG<100 mg/dl, >150 min/week of moderate intensity physical activity, BMI<25 kg/m2, never used tobacco or quit >6 months ago and a healthy diet score),
2. between group mean difference in main risk factors (SBP, DBP, LDL, FPG),
3. proportions meeting >80% of recommended process measures (smoking cessation, moderate or high intensity physical activity, and <5g per person/day salt consumption, >3 daily servings of fruits and vegetables), and 4) proportions achieving or maintaining ten year Framingham CVD risk score15/WHO CVD risk score of <10% or the INTERHEART non-laboratory based score of <5.

Study Intervention Overview:

Usual care arm: The usual care arm will be screened for CVD risk factors. Screening results plus one time education regarding management of risk factors will be provided to all family members. Patients with hypertension, diabetes and dyslipidemia in the control arm will also be referred to primary health care facility. Treatment arm: The study intervention is designed to leverage the existing health care infrastructure available at the community levels. Trained FCHW will be visiting the families to promote lifestyle intervention strategies at least once in two months during the intervention phase.

The intervention consists of three phases: 1) screening and detection of CV risk factors, 2) lifestyle (nutritional/physical activity education and tobacco cessation) counselling 2) FCHW assisted linkage to primary care and 3) active follow-up through a mobile phone application.

Intervention Part 1. Screening for CV risk factors (CONTROL AND TREATMENT ARMS):

All eligible adults in the selected families will undergo a screening procedure for CVD risk factors. The families will be randomized to either the treatment or control arm. At the start of intervention program, high risk patients in the usual care arm will be referred to the existing primary care system for further management.

Intervention Part 2. Lifestyle Education (TREATMENT ARM):

Lifestyle education intervention: The lifestyle education component of the treatment arm includes a minimum of 9 nutritional/tobacco/physical activity consultations. All study participants within the selected families in the treatment arm will participate in the lifestyle education component. Within 30 days of study enrollment, all participants will complete culturally specific food frequency questionnaires (FFQ) and tobacco use surveys. FCHW will receive training from study staff prior to study implementation. Recommended diet modifications for participants will focus on maintaining a healthy weight via redistribution/reduction of calories (by avoiding fried foods and sugar-sweetened beverages), increasing fiber and protein intake via wheat, and sprouted pulses, reducing glycaemic load by switching from refined white rice and bread to whole wheat, increasing fruits and vegetables consumption, and reducing salt and sugar intake. Tobacco cessation and strategies to change the sedentary behaviour will also be discussed in education meetings. Current tobacco users will complete culturally appropriate cessation action guides that identify triggers and action steps to promote tobacco-free behaviours. Family consultations will be repeated after once in every two months to re-assess dietary and tobacco use changes. FCHW workers will conduct peer-support group education meetings with groups of 10 participants once in every two months. Support group meetings will review diet modification and tobacco cessation recommendations and highlight peers' strategies that have led to successful improvement in diet. All individuals with elevated risk factors of CVD will be invited to participate in at least 3 such peer-support group education during the period of the trial.

Intervention Part 3. Linkage to primary care (TREATMENT ARM):

All high risk patients from treatment arm will be linked to appropriate primary care clinics with assistance from FCHW. FCHW workers will assist high risk patients to identify primary or secondary care facilities and will help schedule initial appointments. For 24 consecutive months following initial screening and randomization, participants from intervention arm will receive quarterly phone interviews to measure primary care clinic utilization and to assess cardiovascular risk factor management activities (lipids examined, smoking cessation programs, hypertension control, glucose monitoring).

Care coordination and follow-up:

Each families, in the treatment arm will be assigned a FCHW. During the intervention phase FCHW workers will meet with study patients once in two months to assess study progress and participation in the initial six months. During intermediate-term follow-up (months 7-24) FCHW will maintain once in three months contact with all families. In addition, questionnaire data collection and blood draws at home visits after study months 12 and 24 will help to assess detailed attributes of cardiovascular management (FBG, BP, and LDL measures). An incentivized (free SMS credits) didactic mobile phone SMS platform will be used to enhance follow-up. Via SMS, patients will receive study visit reminders and brief surveys.

Cost effectiveness and acceptability analyses (Aim 3):

The intervention costs will include the resource inputs (e.g., personnel salaries, and materials) that are required to deliver the intervention (in total and per participant). Direct and indirect costs incurred by each family will be estimated using questionnaires. Questionnaires (administered at study visits 0, 12 and 24) will capture direct medical costs, direct non-medical costs (travel), and indirect costs (missed work time, and lost productivity). To estimate the cost-effectiveness (cost per one count decrease in clustering of risk factors), the between trial group difference in intervention delivery and patient direct costs will be divided by the between group difference in clustering of risk factors or cardiovascular risk score: [costs treatment arm - costs standard arm]/[ΣΔPrimary outcome-Treatment arm] - [ΣΔPrimary outcome-usual care arm]. Similarly, incremental cost utility ratio will be calculated using data from a 12 monthly health utility assessment. Quality adjusted life years (QALY) will be used as the measure of health utility.

The acceptability of the interventions will be assessed through qualitative research. Semi-structured FGDs (6 each in men and women) will be conducted among study participants at the end of the intervention period. In-depth interviews with FCHW (6 interviews) will be also conducted to gauge the acceptability of the interventions.

ELIGIBILITY:
Inclusion Criteria:Potential participants must be either parents, children or brothers and sisters of the affected person (individual with documented history of CHD).

More than 18 years of age.

-

Exclusion Criteria:

Bedridden and terminally ill patients. Those who are not willing to provide written informed consent will be also excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1678 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
Composite outcome of multiple cardiovascular risk factors | 2 year
  Proportions achieving blood pressure<140/90 mmHg, fasting blood glucose (FPG)<110 mg/dl, low-density lipoprotein (LDL)<100 mg/dl, and abstinence from smoking/tobacco use.

SECONDARY OUTCOMES:
Blood pressure | 2 year
  Proportion achieving blood pressure<120/80 mmHg, and change in mean systolic and diastolic blood pressure
Blood lipids | 2 Year
  Proportion achieving Total Cholesterol<200 mg/dl and change in mean total cholesterol.
Blood Glucose | 2 year
  Proportion achieving fasting blood glucose<110 mg/dl and change mean fasting blood glucose
Behavioural factors | 2 Year
  >150 min/week of moderate intensity physical activity as assessed from Global Physical Activity Questionnaire , never use of tobacco or quit >6 months ago from structured questionnaire validated by urinary cotinine assessment and a healthy diet score from structured questionnaire.
Acute Coronary Syndrome | 2 year
  Hospital admission for acute coronary syndrome (>24 hours of admission)

CONTACTS AND LOCATIONS:
Overall Officials: Panniyammakal Jeemon, Ph.D, Principal Investigator — Public Health Foundation of India
Locations (1):
- Sree Chitra Tirunal Institute for Medical Sciences and Technology, Trivandrum, Kerala, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jeemon P, Athira T, Lekha TR, Ismail S, Ganapathi S, Harikrishnan S. Family-based interventions for optimal blood pressure outcomes in adults: a cluster randomised controlled trial in India. J Hypertens. 2025 Nov 1;43(11):1871-1877. doi: 10.1097/HJH.0000000000004132. Epub 2025 Sep 3. PMID 40990535
- [Derived] John AS, Ganapathi S, Harikrishnan S, Lekha TR, Stanley A, Soman B, Anish TS, Hadaye R, Cherian JJ, Tandon N, Prabhakaran D, Jeemon P. Within-Trial Cost-Effectiveness Analysis of a Family-Based Structured Lifestyle Modification Intervention Program for Cardiovascular Risk Reduction: Results from the PROLIFIC Trial. Glob Heart. 2025 Jul 31;20(1):65. doi: 10.5334/gh.1450. eCollection 2025. PMID 40757252
- [Derived] Panniyammakal J, Stanley A, Ismail S, Lekha TR, Ganapathi S, Harikrishnan S. Family-Based Interventions to Promote Weight Management in Adults: Results From a Cluster Randomized Controlled Trial in India. Ann Fam Med. 2025 Mar 24;23(2):93-99. doi: 10.1370/afm.230632. PMID 40127979
- [Derived] Jeemon P, Harikrishnan S, Ganapathi S, Sivasankaran S, Binukumar B, Padmanabhan S, Tandon N, Prabhakaran D. Efficacy of a family-based cardiovascular risk reduction intervention in individuals with a family history of premature coronary heart disease in India (PROLIFIC): an open-label, single-centre, cluster randomised controlled trial. Lancet Glob Health. 2021 Oct;9(10):e1442-e1450. doi: 10.1016/S2214-109X(21)00319-3. PMID 34534488
- [Derived] Jeemon P, Harikrishnan S, Sanjay G, Sivasubramonian S, Lekha TR, Padmanabhan S, Tandon N, Prabhakaran D. A PROgramme of Lifestyle Intervention in Families for Cardiovascular risk reduction (PROLIFIC Study): design and rationale of a family based randomized controlled trial in individuals with family history of premature coronary heart disease. BMC Public Health. 2017 Jan 5;17(1):10. doi: 10.1186/s12889-016-3928-6. PMID 28056897